CLINICAL TRIAL: NCT04162171
Title: Noninvasive Cardiac Radioablation for Ventricular Tachycardia
Brief Title: Cohort Study - SBRT for VT Radioablation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: John Sapp (Other)
Responsible Party: Sponsor-Investigator, John Sapp, Staff Physician, Division of Cardiology, Nova Scotia Health Authority
Organization: Nova Scotia Health Authority (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sapp007
Record Dates: First submitted 2019-10-29; First posted 2019-11-14 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Ventricular Tachycardia; Myocardial Infarction; Heart Disease Structural Disorder
MeSH Terms: conditions — Tachycardia, Ventricular; Myocardial Infarction | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Imaging & SBRT Treatment for Ventricular Tachycardia (Experimental)
  Interventions: Radiation: Stereotactic Body Radiotherapy (SBRT) ablation of VT

INTERVENTIONS:
Radiation: Stereotactic Body Radiotherapy (SBRT) ablation of VT — Additional imaging for SBRT planning and implementation:
  * Planning CT (pCT) - CT simulator that utilizes a respiratory positioning monitoring (RPM) optical tracking system and SBRT immobilization setup to provide necessary data to allow for monitoring of the patient's deep inspiration breath-hold (DIGH) maneuver during treatment delivery.
  * SBRT treatment - 30 min procedure on a TrueBeam 1 linear accelerator using SBRT fixation. Patient alignment and DIBH maneuver from the pCT will be replicated using the on-board cone-beam CT (CBCT) guidance and RPM systems.
  Other Names: VT Radioablation

SUMMARY:
Ventricular tachycardia (VT) contributes to over 350,000 sudden deaths each year in the US. Malignant VTs involve an electrical "short circuit" in the heart, formed by narrow channels of surviving tissue inside myocardial scar. Current treatment for VT consists of either implantable defibrillators (ICDs), suppressive drug therapy, catheter ablation or a combination of all 3.

Implantable Defibrillators (ICDs) reduce sudden death and can terminate some ventricular tachycardia (VT) without shocks, but they don't prevent VT. The occurrence of ≥1 ICD shock is associated with reductions in mental well-being and physical functioning, and increases in anxiety and sometimes depression. Further, ICD shocks have been consistently associated with adverse outcomes, including heart failure and death. Furthermore, the most important predictor of ICD shocks is a history of prior ICD shocks.

Therapies to suppress VT include antiarrhythmic drug therapy and catheter ablation, neither however is universally effective. When VT recurs despite antiarrhythmic drug therapy and catheter ablation, novel yet invasive, approaches may be required. Such invasive procedures carry consequent risks of cardiac and extra-cardiac injury.

Stereotactic body radiotherapy (SBRT) is a non-invasive technique that delivers high doses of radiation precisely to specified regions in the body, while minimizing exposure to adjacent tissue. This technique is currently, and commonly used in the treatment of cancer. Conventional application of SBRT has made use of its ability to spare non-target tissue, including for treatment of tumors near the heart. More recently, clinicians have changed the paradigm, by focusing radioablative energy on ventricular scar responsible for ventricular tachycardia. Pre-clinical studies have supported the concept and were followed by first-in-human VT therapeutic experience in 2017. Subsequent studies have had encouraging results for patients who failed or were unable to tolerate conventional treatment.

DETAILED DESCRIPTION:
This will be a single centre single arm prospective cohort study. 12 patients with ventricular tachycardia will be recruited from those who have failed or were unable to tolerate conventional therapy. These patients will be recruited from the cardiology clinic where they will already be under the care of a heart rhythm/heart function specialist. Clinical imaging data, medical history and previous ablation data will be collected and use towards planning their treatment with SBRT. Patients will undergo further imaging (unless recently done clinically), including: 4D cardiac CT (cCT), cardiac MRI (cMRI) and a planning CT (pCT). MRIs will only be performed on patients with ICDs for whom it is considered safe to do so. Using the imaging and electroanatomic substrate mapping data collected from a previous ablation attempt, a volumetric modulated arc therapy (VMAT) treatment plan will be established. This treatment plan will be generated in consultation between the cardiac electrophysiologist, radiation oncologist and medical physicist; and will define the target volume (TV) of myocardial tissue to be treated.

Once a TV has been established and verified, patients will be set up on a TrueBeam 1 linear accelerator where the treatment will be administered. The actual time for treatment administration is approximately 30 minutes.

After the procedure, at 6 & 12 weeks, 7.5 months then every 6 months, a follow-up will occur as a part of standard care where outcome data regarding the chronic success of the ablation procedure will be collected and ICD interrogation will be performed. No imaging or mapping is planned at the follow-up. Patients will be followed for a minimum of 7.5 months to a maximum of 2 years depending on when they are enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Structural heart disease: ischemic or non-ischemic cardiomyopathy diagnosed with cardiac imaging demonstrating either segmental myocardial dysfunction, or presence of scar, AND
* One of the following monomorphic VT events despite prior attempted catheter ablation (or contraindication for ablation), AND despite treatment with a class III antiarrhythmic drug (contraindicated, ineffective or not tolerated): A: Documented sustained monomorphic VT terminated by pharmacologic means, DC cardioversion or manual ICD Therapy. B: ≥3 episodes of monomorphic VT treated with antitachycardia pacing (ATP), at least one of which was symptomatic C: ≥ 5 episodes of monomorphic VT treated with antitachycardia pacing (ATP) regardless of symptoms D: ≥1 appropriate ICD shocks, E: ≥3 monomorphic VT episodes within 24 hours ** VT events must be confirmed by ECG/monitor or ICD download.

Exclusion Criteria:

* Unable or unwilling to provide informed consent
* Have received prior radiotherapy to the likely treatment field
* Inotrope-dependent heart failure or an anticipated life-expectancy of < 1 year in the absence of VT
* Presenting arrhythmia: polymorphic VT or ventricular fibrillation (VF)
* Pregnancy
* Active ischemia (acute thrombus diagnosed by coronary angiography, or dynamic ST segment changes demonstrated on ECG) or another reversible cause of VT (e.g. drug-induced arrhythmia), had recent acute coronary syndrome within 30 days thought to be due to acute coronary arterial thrombosis, or have CCS functional class IV angina. Note that biomarker level elevation alone after ventricular arrhythmias does not denote acute coronary syndrome or active ischemia.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Comparative analysis of ventricular arrhythmia events | During the first 6 months post blanking period vs. 6 months prior to treatment.
  Number of patients with a reduction in the absolute number of ventricular arrhythmia events following ablation and blanking period, in comparison with those prior to treatment.
Comparative analysis of targeting methods assessed by volume of sparred healthy tissue | From time of enrollment to 7.5 ,months post treatment.
  Effectiveness of different myocardial substrate targeting methods on sparing non-target tissue. Delivered treatment approach as compared to a proposed calculated treatment plan using a single phase of the 4DcCT. Measured differences between 2 target-method volumes will equate to the volume of sparred tissue.

SECONDARY OUTCOMES:
Number of patients with procedural complications, including: all cause mortality, pericarditis, pneumonitis, heart failure hospitalization and extra-cardiac injury | Through study completion,min of 7.5 months to max of 2 years.
  Composite of; all cause mortality, pericarditis, pneumonitis, heart failure hospitalization and extra-cardiac injury.
Time to Recurrent Arrhythmia Outcomes | Through study completion,min of 7.5 months to max of 2 years
  Composite of; appropriate ICD shock, VT storm, incessant VT, sustained VT below ICD detection and appropriate antitachycardia pacing.
Ventricular arrhythmia Burden | During 6 months prior vs. 6 months following treatment.
  Composite of; number of appropriate shocks, number of inappropriate shocks, number of antitachycardia pacing events.

CONTACTS AND LOCATIONS:
Overall Officials: John Sapp, MD FRCPC, Principal Investigator — Nova Scotia Health Authority; James Clarke, MD FRCPC, Study Director — Nova Scotia Health Authority; James Robar, Phd FCCPM, Study Director — Nova Scotia Health Authority; Jean-Philippe Pignol, MD FRCPC, Study Director — Nova Scotia Health Authority
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: No